CLINICAL TRIAL: NCT06252363
Title: Knowledge, Practices, and Acceptance of Physiotherapists About the Use of Immersive Virtual Reality in Clinical Practice: An International Online Survey.
Brief Title: Knowledge, Practices, and Acceptance of Physiotherapists About the Use of Immersive Virtual Reality in Clinical Practice.
Status: Completed | Type: Observational
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Other Study IDs: VR-PHYSIO
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Immersive Virtual Reality
Keywords: Physiotherapy; Physical Therapy; Survey; Clinical practice

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Practicing physiotherapists: French- or Dutch-speaking physiotherapists currently practicing their profession

SUMMARY:
Objective: The aim of this online cross-sectional survey is to investigate the knowledge, practices, and acceptance of use of immersive virtual reality (VR) in clinical practice in physiotherapists.

Methods: Physiotherapists from different French-speaking and Dutch-speaking countries will be recruited using non-probability sampling. The survey will be available online on LimeSurvey software for a period of 4 months. The questionnaire will include questions about: general data; knowledge about immersive VR; immersive VR usage in clinical practice; intention to use immersive VR; attitudes towards immersive VR; perceived usefulness of immersive VR; perceived ease of use of immersive VR; social influence on using immersive VR.

Discussion: This study will be the first to investigate the knowledge, practices, and acceptance of use of immersive VR in clinical practice in physiotherapists from different countries around the world. This investigation could lead to a better understanding of the current (non-)implementation of this means of rehabilitation in physiotherapy, and help develop ways to better implement it in physiotherapists' clinical practice.

DETAILED DESCRIPTION:
Background: For several years now, the use of immersive virtual reality (VR) has been studied as an intervention in physiotherapy. This new means of rehabilitation, which can be used not only in hospitals but also at home and in private practice, is promising and appears to be as effective as established treatments. Although the number of studies demonstrating the effectiveness of immersive VR in physiotherapy is growing, its implementation in clinical practice remains relatively low. At present, we do not know the reasons for the lack of use of immersive VR in clinical practice among physiotherapists. Various hypotheses could be envisaged, such as a lack of knowledge or negative attitudes towards it. Conversely, we don't know the exact reasons why some physiotherapists decided to use immersive VR in their clinical routine.

Objective: The aim of this online cross-sectional survey is to investigate the knowledge, practices, and acceptance of use of immersive VR in clinical practice in physiotherapists.

Methods: Physiotherapists from different French-speaking and Dutch-speaking countries will be recruited using non-probability sampling. The survey will be available online on LimeSurvey software for a period of 4 months. The questionnaire will include questions about: general data; knowledge about immersive VR; immersive VR usage in clinical practice; intention to use immersive VR; attitudes towards immersive VR; perceived usefulness of immersive VR; perceived ease of use of immersive VR; social influence on using immersive VR.

Discussion: This study will be the first to investigate the knowledge, practices, and acceptance of use of immersive VR in clinical practice in physiotherapists from different countries around the world. This investigation could lead to a better understanding of the current (non-)implementation of this means of rehabilitation in physiotherapy, and help develop ways to better implement it in physiotherapists' clinical practice.

ELIGIBILITY:
Eligibility Criteria:

* To have a degree in physiotherapy
* Currently practicing as a physiotherapist
* To speak French or Dutch

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: French-speaking or Dutch-speaking graduates in physiotherapy currently practicing as physiotherapists.
Sampling Method: Non-Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2024-02-23 (Actual); Primary Completion 2024-07-23 (Actual); Study Completion 2024-07-23 (Actual)

PRIMARY OUTCOMES:
Knowledge about immersive virtual reality | Baseline (at the time of completing the questionnaire)
  General knowledge about immersive virtual reality will be assessed using closed questions.
Use of immersive virtual reality (practice) | Baseline (at the time of completing the questionnaire)
  Use of immersive virtual reality will be assessed using closed questions (e.g., duration and frequency of use, pathologies treated, age of patients treated, system used, type of rehabilitation,...).
Intention to use immersive virtual reality | Baseline (at the time of completing the questionnaire)
  Intention to use immersive virtual reality will be assessed using closed questions (e.g., research performed by oneself, readiness to invest,...).
Attitudes towards immersive virtual reality | Baseline (at the time of completing the questionnaire)
  Attitudes towards immersive virtual reality will be assessed using Likert-scale questions (e.g., desire to find out more, perceived suitability for different people,...).
Perceived usefulness of immersive virtual reality | Baseline (at the time of completing the questionnaire)
  Perceived usefulness of immersive virtual reality will be assessed using Likert-scale questions (e.g., general usefulness in physiotherapy, usefulness for different clinical outcomes, usefulness as a means of rehabilitation,...).
Perceived ease of use of immersive virtual reality | Baseline (at the time of completing the questionnaire)
  Perceived ease of use of immersive virtual reality will be assessed using Likert-scale questions (ease of use for oneself, patients, and other physiotherapists).
Social influence on using immersive virtual reality | Baseline (at the time of completing the questionnaire)
  Social influence on using immersive virtual reality will be assessed using Likert-scale questions (influence of people inside and outside the workplace on using immersive virtual reality in clinical practice).

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Pitance, PhD, Principal Investigator — Université Catholique de Louvain
Locations (1):
- Université Catholique de Louvain, Brussels, Belgium